CLINICAL TRIAL: NCT03763851
Title: Cannabis Oil and Radiation Therapy for the Management of Pain: Assessment of Safety and Efficacy in a Randomized, Double-blind Placebo-controlled Phase II/III Clinical Trial
Brief Title: Cannabis Oil and Radiation Therapy for the Management of Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to mycotoxin potential contamination of one lot of study drug
Sponsor: Tetra Bio-Pharma (Industry)
Collaborators: Santé Cannabis (Other); McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPP005-Ph2/3-01
Record Dates: First submitted 2018-11-12; First posted 2018-12-04 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Prostate Cancer; Lung Cancer; Breast Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Lung Neoplasms; Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabis group (Experimental): Delta-9 Tetrahydrocannabidiol (THC) /Cannabidiol (CBD) ratio 1:1 capsule
  These capsules contain different cannabis formulations with low-dose and high-dose preparations according to the treatment group:
  * Cannabis group low-dose capsule contains THC 1mg CBD 1mg
  * Cannabis group high-dose capsule contains THC 2.5mg CBD 2.5mg
  Interventions: Radiation: Active PPP005; Radiation: Radiotherapy
- Placebo group (Placebo Comparator): The placebo capsule will have no cannabis, it will look identical to the active treatment capsule, and it will also be prepared in "low-dose" and "high-dose" presentations.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Active PPP005 — Group assigned to active PPP005 in the randomized placebo-controlled trial
  Arms: Cannabis group
Radiation: Radiotherapy — Palliative RadioTherapy to the symptomatic site

SUMMARY:
In this innovative approach seeking effective therapeutic strategies, the investigators are proposing to test the effectiveness of medical cannabis oil as an adjunct to palliative Radiation Therapy (RT) and Best Supportive Care to alleviate cancer pain that was only partially relieved with conventional medications. Furthermore, the investigators will assess the effect of medical cannabis oil on health-related quality of life and symptoms that are frequently associated with metastatic cancers including fatigue, anxiety, depression, insomnia and decreased appetite. The safety profile of medical cannabis oil with respect to prolonged use of more than two weeks of administration, concomitant medication use and palliative RT will also be examined.

DETAILED DESCRIPTION:
This is a 6-week randomized, double-blind, placebo-controlled, parallel group design trial followed by an open-label extension phase of 12 weeks, to evaluate tolerability of medical cannabis oil to reduce chronic pain intensity.

Consecutive adult patients between the ages of 18 and 75, male and female, with cancer pain, with an average weekly pain intensity score greater than 4 on the 11 points Numerical Rate Scale (NRS), will be prospectively recruited and invited to participate in this trial.

Informed consent will be obtained by a Research Assistant.

After baseline documentation with standardized scales, patients will be randomized to one of two parallel groups:

* Cannabis group: Delta-9 Tetrahydrocannabidiol (THC) /Cannabidiol (CBD) ratio 1:1 capsule
* Placebo group: Placebo capsule
* All patients will receive palliative RT to the symptomatic site. Patients will have a dose titration phase during the first week. The dose escalation will allow patients to adapt to the potential adverse effects (AEs) of the medical cannabis.

Follow-up visits either in person or by phone will be at 1 week, 3 weeks and 6 weeks of treatment.

At the end of the first phase of the study, patients who wish to participate in the open-label extension phase will have the option to continue in the same treatment regimen. For the placebo group, patients will have the option to receive the active treatment during the 12-week open-label phase if the study physician feels it may potentially provide benefits. Similarly, the dose will be titrated up in the placebo group who wants to receive the active drug in the extension program.

The open-label phase is 12 weeks long. For this open-label extension phase the follow-up visits will be done after 4 weeks and 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to consent to the study-specific written consent form, in English or French;
2. Adult patients, male and female between the ages of 18 and 75 (inclusively);
3. Patients with confirmed diagnosis of metastatic carcinoma of the prostate, lung or breast;

   1. No limitation with respect to number of metastases (bone and visceral);
   2. Location of metastases limited to exclude any brain metastases
4. Patients experiencing an average weekly pain intensity score of 4 or higher on a 11 points NRS and requiring palliative RT;
5. KPS of equal or higher than 60;
6. Subject agreed to follow the protocol;
7. Patients who are referred to receive RT and are non-regular users of cannabis in any form (three times per week or more) and are willing to abstain for 1 week prior and during the study;
8. Patients receiving opioids and other concomitant pain medications must have a stable dose for the last 15 days;
9. Normal cognitive status according to MiniCog;
10. Normal liver function (defined as aspartate aminotransferase 10-40 U/L and alanine aminotransferase 7-56 U/L)
11. Normal renal function (defined as serum creatinine level <133 µmol/L and Estimated Glomerular Filtration Rate (eGFR) equal or higher than 60)
12. Negative result on βhuman chorionic gonadotropin pregnancy test (if applicable)
13. A female volunteer must meet one of the following criteria:

    1. If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first drug administration, during the study and for at least 60 days after the last dose.
    2. If of non-childbearing potential - should be surgically sterile or in a menopausal state
14. A male volunteer with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must be surgically sterile or agrees to use one of the accepted contraceptive regimens from first drug administration until 3 months after the last drug administration.

Exclusion Criteria:

1. Patients who are unable to consent or to comply with the instructions of the study;
2. Patients suffering primarily from pain not related to cancer;
3. KPS of < 60;
4. Previous serious adverse event or hypersensitivity to cannabis or cannabinoids;
5. Presence of significant cardiac disease (history of unstable ischemic heart disease, heart failure, severe and uncontrolled hypertension) that, in the opinion of the investigator, would put the patient at risk of a clinically significant arrhythmia or myocardial infarction;
6. Current substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM 5);
7. Life-time history of dependence on cannabis or diagnosis of cannabis use disorder (CUD) according to the DSM 5;
8. Life-time history of DSM 5 schizophrenia, bipolar disorder, or previous psychosis with or intolerance to cannabinoids;
9. Current suicidal ideation according to the Columbia-Suicide Severity Rating Scale (C-SSRS);
10. Pregnant, breast-feeding or female patients of child-bearing potential and male patients whose partner is of child-bearing potential, unless willing to ensure that they or their partner use effective contraception;
11. Hepatic impairment (aspartate aminotransferase more than three times normal) or renal function impairment (serum creatinine level >133 µmol/L.
12. Cognitive impairment according to MiniCog;
13. Current use of cannabis in any form more than 3 times per week or use of cannabinoid-based medications within 7 days of study entry and refusal to abstain for the duration of the study;
14. Positive blood test for cannabinoids at screening or positive urine screening for other potential abuse substances (e.g. alcohol, cocaine, amphetamines and methamphetamines, unprescribed opioids);
15. Participation in another clinical trial within 30 days of screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Cancer pain intensity assessed by Pain Intensity (PI) measurement a numerical rating scale | Change (a reduction of 30% in pain intensity) in pain intensity after medical cannabis oil administration compared to placebo at 6 weeks compared to baseline
  Pain Intensity (PI) measurement a Numerical Rating Scale (zero= no pain and 10= pain as bad as it can be).
  A reduction of PI ≥ 33% will be considered as a clinically important level of pain relief
Cancer pain quality using the Brief Pain Inventory-SF (BPI-SF) | The measurements will be completed at baseline before initiating treatment and at week 1, week 3 and week 6 after starting treatment
  The BPI-SF consists of nine questions; eight have a single response, and Question 9 is subdivided into seven parts. The Total BPI for Question 9 is the unweighted sum of the seven assessments and represents the effect of pain

SECONDARY OUTCOMES:
Impact of medical cannabis oil combined with radiation treatment on HRQoL as measured by the EQ-5D-5L | at baseline, 1-week, 3-week, and 6-week follow-up
Functional status assessed by the Functional Assessment of Cancer Therapy for Prostate patients (FACT-P). | The measurements will be completed at baseline before initiating treatment and at week 1, week 3 and week 6 after starting treatment
Fatigue burden assessed by the Brief Fatigue Inventory (BFI). | The measurements will be completed at baseline before initiating treatment and at week 1, week 3 and week 6 after starting treatment
Cognitive status assessed by the Mini-Cog | The measurements will be completed at baseline before initiating treatment and at week 1, week 3 and week 6 after starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Niazi, MD, Principal Investigator — Jewish General Hospital, McGill University; Jean Zigby, MD, Principal Investigator — Jewish General Hospital, McGill University
Locations (1):
- Sante Cannabis, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided